CLINICAL TRIAL: NCT06974955
Title: A Real-World, Multicenter, Retrospective Study to Evaluate the Clinical Performance and Safety of MantraTM Surgical Robotic System for Soft Tissue Surgeries
Brief Title: A Study on the Safety and Effectiveness of the Mantra™ Surgical Robotic System for Soft Tissue Surgeries
Acronym: MARS
Status: Not yet recruiting | Type: Observational
Sponsor: Sudhir Srivastava Innovations Pvt. Ltd. (Industry)
Collaborators: Clicebo Solutions Private Limited (Other)
Responsible Party: Sponsor
Other Study IDs: CSPL/REG/2025/01
Record Dates: First submitted 2025-04-03; First posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Soft Tissue Surgeries
Keywords: Retrospective Study; Real World; Mantra TM Surgical Robotic System; soft tissue surgeries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients who have previously undergone surgery using the Mantra™ Surgical Robotic System 3.0

SUMMARY:
A Real-World, multicentre retrospective study to evaluate the clinical performance and safety of MantraTM Surgical Robotic System for soft tissue surgeries.

The purpose of this retrospective study is to evaluate the clinical performance and safety of the Mantra™ Surgical Robotic System, Model 3.0, for soft tissue surgeries. It aims to provide real-world evidence on the system's reliability, safety, and effectiveness in the real world population. The SSI Mantra 3.0 Surgical Robotic System is an advanced, modular, and cost-effective robotic-assisted surgical platform designed to enhance precision, flexibility, and control in minimally invasive surgeries (MIS).

The objective of this retrospective study is to assess the clinical performance and safety of the Mantra™ Surgical Robotic System in performing various soft tissue surgeries based on retrospective data analysis.

DETAILED DESCRIPTION:
A Real-World, multicentre retrospective study to evaluate the clinical performance and safety of MantraTM Surgical Robotic System for soft tissue surgeries.

Objective : To assess the clinical performance and safety of the Mantra™ Surgical Robotic System in performing various soft tissue surgeries based on retrospective data analysis.

Study Outcomes: The retrospective analysis of the Mantra Surgical Robotic System focused on evaluating its clinical performance, safety and efficacy in minimally invasive surgeries. The study outcomes were assessed based on surgical safety and efficacy parameters, intraoperative efficiency, post-operative recovery, and system utilization trends.

Primary Study Outcomes

1. Primary Effectiveness Endpoint

   * Rate of Unplanned Conversion to other minimally invasive surgery (MAS) or open surgery (OP).
   * Successful completion of the procedure using the SSI Mantra 3.0 Surgical Robotic System as planned.
2. Primary Safety Endpoint

   * Rate of Total Intraoperative and Postoperative Serious Adverse Events (SAE) up to 30 days post-procedure.
   * Assessment of device-related complications . Secondary Study Outcomes

1. Operative Time

* Measured from skin incision to skin closure to assess efficiency. 2. Estimated Blood Loss (Intraoperative)
* Quantification of blood loss during surgery. 3. Need for Blood Transfusion
* Evaluation of cases requiring intraoperative blood transfusion. 4. Intraoperative Complications
* Identification and classification of adverse events occurring during surgery. 5. Return to Operating Room within 24 Hours
* Evaluation of unplanned reoperations. 6. Length of Hospital Stay
* Time from hospital admission to discharge post-surgery. 7. Readmission to Hospital within 30 Days
* Tracking of unexpected hospital readmissions. 8. Reoperation within 30 Days
* Incidence of repeat surgical interventions. 9. Mortality Rate at 30 Days
* Evaluation of patient survival post-procedure. 10. Device Deficiencies and Use Errors
* Documentation of device-related malfunctions or improper usage. 11. All Adverse Events
* Comprehensive assessment of both minor and major adverse effects. 12. Device Performance Data
* Monitoring of unplanned instrument usage, system clashes, collision detection, and alarm activations.

Timepoints: Day of surgery - 30 days (follow-up). Study Design: This is a retrospective, multicentre study designed to collect and analyze data from surgeries performed using the Mantra™ Surgical Robotic System, Models 3.0,. The study will evaluate clinical performance, safety, and patient outcomes across approximately twenty centers with a target sample size of 365 patients.

ELIGIBILITY:
Inclusion Criteria:

- Participants must meet all of the following criteria to be eligible for inclusion in this retrospective clinical study of the SSI Mantra 3.0 Surgical Robotic System.

Patients who have previously undergone surgery using the Mantra™ Surgical Robotic System (Model 3.0) for the following procedures mentioned in Appendix D

Exclusion Criteria:

* Patients with missing data on primary endpoints.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will include patients who have undergone soft tissue surgeries using the Mantra™ Surgical Robotic System (3.0)
Sampling Method: Non-Probability Sample
Enrollment: 365 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Rate of Unplanned Conversion to other minimally invasive surgery (MAS) or open surgery (OP) | 1 day
  • Rate of Unplanned Conversion to other minimally invasive surgery (MAS) or open surgery (OP).
Successful completion of procedures without the need for conversion | 1 day
  Successful completion of procedures without the need for conversion
Rate of intraoperative and postoperative serious adverse events (SAEs) occurring up to 30 days post-procedure | 30 days
  Rate of intraoperative and postoperative serious adverse events (SAEs) occurring up to 30 days post-procedure
Evaluation of surgical complications, including infections, haemorrhage, and device-related adverse events | 30 day
  Evaluation of surgical complications, including infections, haemorrhage, and device-related adverse events

SECONDARY OUTCOMES:
Operative Time - Measured from skin incision to skin closure to assess efficiency | 1 day
  Measured from skin incision to skin closure to assess efficiency
Estimated Blood Loss (Intraoperative) - Quantification of Blood loss during surgery | 1 day
  Quantification of blood loss during surgery
Need for Blood Transfusion - Evaluation of cases requiring intraoperative blood transfusion | 1 day
  Evaluation of cases requiring intraoperative blood transfusion
Intraoperative Complications - Identification and classification of adverse events occurring during surgery | 1 day
  Identification and classification of adverse events occurring during surgery
Return to Operating Room within 24 Hours - Evaluation of unplanned reoperations | 1 day
  Evaluation of unplanned reoperations
Length of Hospital Stay - Time from hospital admission to discharge post-surgery | 30 days
  Time from hospital admission to discharge post-surgery
Readmission to Hospital within 30 Days - Tracking of unexpected hospital readmissions | 30 days
  Tracking of unexpected hospital readmissions
Reoperation within 30 Days - Incidence of repeat surgical interventions | 30 days
  Incidence of repeat surgical interventions
Mortality Rate at 30 Days - Evaluation of patient survival post-procedure | 30 days
  Evaluation of patient survival post-procedure
Device Deficiencies and Use Errors - Documentation of device-related malfunctions or improper usage | 1 day
  Documentation of device-related malfunctions or improper usage
All Adverse Events - Monitoring of all minor and major adverse events related to surgery | 30 days
  Monitoring of all minor and major adverse events related to surgery
Device Performance Metrics - Assessment of unplanned instrument usage, robotic arm clashes, collision detection, and system-generated alarms | 1 day
  Assessment of unplanned instrument usage, robotic arm clashes, collision detection, and system-generated alarms

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Dr. Somashekhar S P, MBBS, MS, MCh, FRCS, FRCS, Principal Investigator — Aster CMI Hospital
Locations (1):
- ASTER CMI Hospital, Bangalore, Karnataka, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stoianovici DC, Patriciu A, Mazilu D, et al. AcuBot: a robot for radiological interventions. IEEE Trans Rob Autom. 2003; 19: 926-30.
- [Background] Gomez G. Sabiston Textbook of Surgery. 17th ed. Philadelphia, Pa: Elsevier Saunders; 2004. Emerging Technology in surgery: informatics, electronics, robotics.
- [Background] US Food and Drug Administration. Use of real-world evidence to support regulatory decision-making for medical devices: guidance for industry and Food and Drug Administration staff. Food and Drug Administration. 2017 Aug 31
- [Background] Hutchinson A. The top 50 inventions of the past 50 years. Popular Mechanics. December 2005.
- [Background] Boctor EM, Choti MA, Burdette EC, Webster Iii RJ. Three-dimensional ultrasound-guided robotic needle placement: an experimental evaluation. Int J Med Robot. 2008 Jun;4(2):180-91. doi: 10.1002/rcs.184. PMID 18433079
- [Background] Cadeddu JA, Bzostek A, Schreiner S, Barnes AC, Roberts WW, Anderson JH, Taylor RH, Kavoussi LR. A robotic system for percutaneous renal access. J Urol. 1997 Oct;158(4):1589-93. PMID 9302179
- [Background] Harris SJ, Arambula-Cosio F, Mei Q, Hibberd RD, Davies BL, Wickham JE, Nathan MS, Kundu B. The Probot--an active robot for prostate resection. Proc Inst Mech Eng H. 1997;211(4):317-25. doi: 10.1243/0954411971534449. PMID 9330543
- [Background] Tan GY, Goel RK, Kaouk JH, Tewari AK. Technological advances in robotic-assisted laparoscopic surgery. Urol Clin North Am. 2009 May;36(2):237-49, ix. doi: 10.1016/j.ucl.2009.02.010. PMID 19406324
- [Background] Kazanzides P, Fichtinger G, Hager GD, Okamura AM, Whitcomb LL, Taylor RH. Surgical and Interventional Robotics: Core Concepts, Technology, and Design. IEEE Robot Autom Mag. 2008 Jun 1;15(2):122-130. doi: 10.1109/MRA.2008.926390. No abstract available. PMID 20428333
- [Background] Sim HG, Yip SK, Cheng CW. Equipment and technology in surgical robotics. World J Urol. 2006 Jun;24(2):128-35. doi: 10.1007/s00345-006-0070-6. Epub 2006 Mar 15. PMID 16538515
- [Background] H. Lavery, D. Samadi, and A. Levinson, "Not a zerosum game: the adoption of robotics has increased overall prostatectomy utilization in the united states," in Proceedings of the American Urological Association Annual Meeting, Poster Session,Washington, DC, USA, 2011.
- [Background] Hashizume M, Tsugawa K. Robotic surgery and cancer: the present state, problems and future vision. Jpn J Clin Oncol. 2004 May;34(5):227-37. doi: 10.1093/jjco/hyh053. PMID 15231856
- [Background] Camarillo DB, Krummel TM, Salisbury JK Jr. Robotic technology in surgery: past, present, and future. Am J Surg. 2004 Oct;188(4A Suppl):2S-15S. doi: 10.1016/j.amjsurg.2004.08.025. PMID 15476646
- [Background] Marohn MR, Hanly EJ. Twenty-first century surgery using twenty-first century technology: surgical robotics. Curr Surg. 2004 Sep-Oct;61(5):466-73. doi: 10.1016/j.cursur.2004.03.009. PMID 15475097
- [Background] Ballantyne GH. The pitfalls of laparoscopic surgery: challenges for robotics and telerobotic surgery. Surg Laparosc Endosc Percutan Tech. 2002 Feb;12(1):1-5. doi: 10.1097/00129689-200202000-00001. PMID 12008756
- See also: Related Info — https://www.intuitive.com/en-us/about-us/company/clinical-evidence
- See also: Related Info — http://www.intuitivesurgical.com/company/regulatory-clearance.html